CLINICAL TRIAL: NCT02082522
Title: Multicenter, Open-label, Randomized, Controlled Phase III Clinical Study of the Efficacy and Safety of Photodynamic Therapy Using Porfimer Sodium for Injection as Treatment for Unresectable Advanced Perihilar Cholangiocarcinoma
Brief Title: Efficacy and Safety Study of PDT Using Photofrin in Unresectable Advanced Perihilar Cholangiocarcinoma (OPUS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual rate remaining too low
Sponsor: Concordia Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIN-PHO1201
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Unresectable perihilar cholangiocarcinoma; Klatskin tumor; Photodynamic therapy; Porfimer sodium; Photofrin; Gemcitabine; Cisplatin; Stents; CCA; PDT; Bile duct cancer; Bile duct tumor; Bile duct adenocarcinoma; Chemotherapy
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Drug Therapy; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photodynamic therapy-Photofrin plus SMC (Experimental): Photodynamic therapy (PDT) involves the i.v. injection of Photofrin followed by the illumination of the tumor using a fiber optic device. Two days after the injection, a laser light (180 J/cm(2)) will be applied to the tumor. A second light application will be given 96-120 hours after Photofrin injection if PDT could not initially be performed on all sides of the tumor. Post illumination, all patients will undergo stenting as part of standard medical care procedure. Up to 3 additional courses of PDT using a light dose of 120 J/cm(2) may be given at 3-month intervals. Standard Medical Care (SMC) is defined as stenting procedure plus chemotherapy regimen.
  Interventions: Drug: Photodynamic therapy-Photofrin; Procedure: Stenting procedure; Drug: Chemotherapy regimen
- Standard Medical Care (SMC) (Active Comparator): Standard Medical Care (SMC) is defined as stenting procedure plus chemotherapy regimen. The chemotherapy regimen will comprise gemcitabine (1 000 mg/m(2)) followed by cisplatin (25 mg/m(2)), each administered on days 1 and 8 every 3 weeks (21 day-cycle) for four cycles. An additional 12 weeks of the same chemotherapy regimen may be administered if there is no disease progression or intolerable toxicity.
  Interventions: Procedure: Stenting procedure; Drug: Chemotherapy regimen

INTERVENTIONS:
Drug: Photodynamic therapy-Photofrin — Photodynamic therapy (PDT) involves the i.v. injection of Photofrin (2 mg/kg) followed by the illumination of the tumor using a fiber optic device during an endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC). Two days after the injection, a laser light (180 J/cm(2)) will be applied to the tumor. A second light application will be given 96-120 hours after Photofrin injection if PDT could not initially be performed on all sides of the tumor. Post illumination, all patients will undergo stenting as part of standard medical care procedure. Up to 3 additional courses of PDT using a light dose of 120 J/cm(2) may be given at 3-month intervals.
  Other Names: PDT-Photofrin
  Arms: Photodynamic therapy-Photofrin plus SMC
Procedure: Stenting procedure — As per standard medical procedures, stenting procedure consists in the placement of stents above the main tumors of the right and left hepatic bile ducts via endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC) when the ERCP approach has been unsuccessful.
  Other Names: Stents placement
Drug: Chemotherapy regimen — The regimen will comprise gemcitabine (1 000 mg/m(2)) followed by cisplatin (25 mg/m(2)), each administered on days 1 and 8 every 3 weeks (21 day-cycle) for four cycles. An additional 12 weeks of the same chemotherapy regimen may be administered if there is no disease progression or intolerable toxicity.
  Other Names: Gemcitabine/Cisplatin

SUMMARY:
Photodynamic therapy (PDT) is a combination of a drug, porfimer sodium (Photofrin), which is activated by a light from a laser that emits no heat. This technique works to allow the medical doctor to specifically target and destroy abnormal or cancer cells while limiting damage to surrounding healthy tissue. The activation of the drug is done by lighting the abnormal areas using a fiber optic device (very fine fiber like a fishing line that permits light transmission) inserted into a flexible tube with a light called cholangioscope for the bile duct. The light will activate the porfimer sodium concentrated in the abnormal tissue, leading to its destruction.

This research study will evaluate the efficacy and safety of PDT with porfimer sodium administered with Standard Medical Care (SMC) compared to SMC alone on the overall survival time of patients with non-operable advanced cholangiocarcinoma, a rare cancer of the bile ducts. It will involve 200 patients across North America and Europe. Other countries may participate if needed. Participation will last at least 18 months.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is a combination of a drug, porfimer sodium (Photofrin), which is activated by a light from a laser that emits no heat. This technique works to allow the medical doctor to specifically target and destroy abnormal or cancer cells while limiting damage to surrounding healthy tissue. The activation of the drug is done by lighting the abnormal areas using a fiber optic device (very fine fiber like a fishing line that permits light transmission) inserted into a flexible tube with a light called cholangioscope for the bile duct. The light will activate the porfimer sodium concentrated in the abnormal tissue, leading to its destruction.

Cholangiocarcinoma (CCA) is defined as primary malignant tumors of the bile ducts. The exact etiology remains unknown. These cancerous tumors block the bile flow and can be intrahepatic (IH) or extrahepatic (EH). The distinction between IH- and EH-CCA has become increasingly important, as the epidemiological features (i.e., incidence and risk factors), the biologic and pathologic characteristics and the clinical course are largely different. Unfortunately, most subjects are found to have metastases or unresectable disease at the time of diagnosis. Median survival for subjects with unresectable perihilar-CCA varies between five and eight months. The one-year survival is 50%, with 20% surviving at two years and 10% at three years. Unresected CCA is a rapidly fatal process with cholangitis being a significant cause of morbidity and mortality in these subjects.

This study was designed to confirm the efficacy of PHOPDT + standard medical care (SMC) defined as stents plus gemcitabine/cisplatin chemotherapy regimen on the overall survival of subjects with unresectable cholestasis perihilar Bismuth type III or IV - tumor TNM stage III or IVa CCA.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 or older
* Diagnosed with radiologically and biopsy or cytology confirmed inoperable perihilar cholangiocarcinoma Bismuth Tumor Stage III/IV
* Non-menopausal or non-sterile female subjects of childbearing potential must have a negative serum beta-HCG and use a medically acceptable form of birth control
* Able to sign an informed consent

Exclusion Criteria:

* Diagnostic of cholangiocarcinoma made more than 45 days prior to randomization
* Cholangiocarcinoma with extra-hepatic metastasis or concurrent non-solid malignancy
* Presence or history of other neoplasms (treated during the last five years prior to study entry) other than carcinoma in situ of the cervix or basal carcinoma of the skin
* Previously received photodynamic therapy for cholangiocarcinoma
* Previously undergone surgical resection of the cholangiocarcinoma
* Previously undergone chemotherapy, brachytherapy, or radiotherapy prior to entering the study
* Previously undergone metal stent insertion
* Porphyria or hypersensitivity to porphyrins (constituents of porfimer sodium), gemcitabine, cisplatin or other platinum-containing compounds
* Presence of infection other than the infection of the bile duct (cholangitis)
* Acute or chronic medical or psychological illnesses that prevent endoscopy procedures
* Abnormal blood test results
* Severe impairment of your kidney or liver function
* Decompensated cirrhosis
* Pregnant or intend to become pregnant, breastfeeding or intend to breast-feed during this study
* Participated in another drug study within 90 days before this one
* Unable or unwilling to complete the follow-up evaluations required for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (31):
- United States (18):
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - Oschner Medical Center, Kenner, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southwestern Regional Medical Center, Inc., Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Center for Digestive Health - AHN ASRI, Pittsburgh, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - CHUM Hôpital St-Luc, Montreal, Quebec
- Germany (5):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Klinikum Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Johann-Wolfgang-Goethe Universität Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen (AöR), Essen, North Rhine-Westphalia
- South Korea (5):
  - Konkuk University Medical Center, Seoul, Gwangjin-gu
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Seoul National University Hospital, Seoul
- UniversitätsSpital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The study was prematurely discontinued meaning only descriptive analyses are possible. It is not feasible to share this sort of data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An independent expert panel acted as central assessors for subjects across all sites. Central assessors prospectively interpreted all abdominal CT and cholangiogram images taken at screening to establish the final diagnosis and to confirm the randomization. Central assessors had the authority to overrule the investigator's diagnosis.
Groups:
- Photodynamic Therapy-Photofrin Plus SMC: Photodynamic therapy (PDT) involved the i.v. injection of Photofrin (2 mg/kg) followed by the illumination of the tumor using a fiber optic device. Two days after the injection, a laser light (180 J/cm(2)) was applied to the tumor. A second light application was given 96-120 hours after Photofrin injection if PDT could not initially be performed on all sides of the tumor. Post illumination, all patients underwent stenting. Up to 3 additional courses of PDT using a light dose of 120 J/cm(2) could be given at 3-month intervals.
  As per SMC, stenting procedure consisted of the placement of stents above the main tumors of the right and left hepatic bile ducts. The chemotherapy regimen comprised gemcitabine (1 000 mg/m(2)) followed by cisplatin (25 mg/m(2)), each administered on days 1 and 8 every 3 weeks (21 day-cycle) for four cycles. An additional 12 weeks of the same chemotherapy regimen could be administered if there was no disease progression or intolerable toxicity.
- Standard Medical Care (SMC): Standard Medical Care (SMC) was defined as stenting procedure plus chemotherapy regimen. The chemotherapy regimen comprised gemcitabine (1 000 mg/m(2)) followed by cisplatin (25 mg/m(2)), each administered on days 1 and 8 every 3 weeks (21 day-cycle) for four cycles. An additional 12 weeks of the same chemotherapy regimen could be administered if there was no disease progression or intolerable toxicity. As per SMC, stenting procedure consisted of the placement of stents above the main tumors of the right and left hepatic bile ducts.
Period: Overall Study
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Started | 15 | 13
Completed | 0 | 0
Not Completed | 15 | 13
Not completed — Sponsor termination | 5 | 3
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Disease progression | 2 | 2
Not completed — Chemotherapy change | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC) | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.84) | 66.6 (7.69) | 64.9 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  South Korea | 5 | 8 | 13
  United States | 9 | 4 | 13
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time
Description: Time from the date of randomization until the date of death or the last date the subject was known to be alive
Time Frame: Up to 26 months
Population: All participants randomized (intent-to-treat population)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 15 | 13
days | 444 [111.0 to NA] — The value cannot be estimated because less than 50% of patients had a documented death by the time of premature study termination. Only 15 patients were enrolled, most did not complete the study and there was 1 death. Impossible to measure this. | 387 [181.0 to NA] — Value cannot be estimated because < 50% of patients had a documented death at time of premature study termination. Only 13 subjects were enrolled, most did not complete the study & there were 0 deaths in the group. Impossible to measure this.

2. Secondary Outcome: Time-to-bilirubin Response
Description: From the date of randomization until the date of first documented bilirubin response
Time Frame: Up to 30 days
Population: Data not collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Best Overall Tumor Response as Measured by the RECIST 1.1 Criteria (Response Evaluation Criteria in Solid Tumors)
Description: From the start of the treatment until disease progression or recurrence the RECIST 1.1 criteria are applied (Response Evaluation Criteria in Solid Tumors)
Time Frame: Up to 26 months
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 9 | 8
percentage of participants | 56 | 75

4. Secondary Outcome: Time-to-tumor Progression
Description: From the date of first documented response until the date that tumor progression was assessed
Time Frame: Up to 26 months
Population: Not collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline on Karnofsky Performance Scale (KPS)
Description: The Karnofsky Performance Scale scores range from 0% to 100%. The lower the Karnofsky score, the worse likelihood of survival. However, the premature termination of the study does not allow for a meaningful analysis of the scale where 100% means no complaints with no evidence of disease, 80% is normal activity with effort and some signs or symptoms of disease.
Time Frame: Baseline, 7 days
Population: At Day 7, all 15 subjects in the PDT +SMC group were analysed and 9/13 in the SMC Alone group were analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 15 | 9
score on a scale | -0.7 (7.99) | 0 (0)

6. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: The Karnofsky Performance Scale (KPS) scores range from 0% to 100%. The lower the Karnofsky score, the worse likelihood of survival. A score of 100% means there are no complaints and no evidence of disease. A score of 80% means there is normal activity with effort and some signs or symptoms of disease. A score of 0% means death.
Time Frame: Baseline, up to 4 weeks
Population: At 4 weeks, 12 subjects in the PDT +SMC group were analysed and 9 in the SMC Alone group were analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 12 | 9
score on a scale | 1.7 (5.77) | 0 (0)

7. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 6
Time Frame: Baseline, 13 weeks
Population: At 13 weeks, 8 subjects in the PDT +SMC group were analysed and 8 in the SMC Alone group were analysed. Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 8 | 8
score on a scale | 0.0 (7.56) | 2.5 (4.63)

8. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 6
Time Frame: Baseline, 16 weeks
Population: At 16 weeks, 9 subjects in the PDT +SMC group were analysed and 9 in the SMC Alone group were analysed. Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 9 | 9
score on a scale | -6.7 (15.00) | 3.3 (5.00)

9. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 5
Time Frame: Baseline, 29 weeks
Population: At 29 weeks, 6 subjects in the PDT +SMC group were analysed and 5 in the SMC Alone group were analysed. Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 6 | 5
score on a scale | 0.0 (8.94) | 2.0 (4.47)

10. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 5
Time Frame: Baseline, 41 weeks
Population: At 41 weeks, 2 subjects in the PDT +SMC group were analysed and 1 in the SMC Alone group was analysed. Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 2 | 1
score on a scale | 10.0 (14.14) | 0.0 (0.0)

11. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 5
Time Frame: Baseline, 54 weeks
Population: At 54 weeks, only 1 subject in each group was measured. Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 1 | 1
score on a scale | 0.0 (0.0) | 0.0 (0.0)

12. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 5
Time Frame: Baseline, 66 weeks
Population: Data not collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Performance Status on the Karnofsky Performance Scale (KPS)
Description: as for outcome 5
Time Frame: Baseline, 78 weeks
Population: Not collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30)
Description: Final European Organisation for Research and Treatment of Cancer (EORTC) scores for multi-item scales and single-item measures will range from 0 to 100. This questionnaire assesses the quality of life of cancer patients. A high score represents a high/healthy level of functioning, basically a high Quality of Life.
Time Frame: Baseline, 7 days
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 15 | 9
score on a scale | -2.2 (30.29) | 0.0 (0.0)

15. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, up to 4 weeks
Population: Not collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 13 weeks
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 7 | 8
score on a scale | -7.1 (30.59) | 6.2 (35.84)

17. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 16 weeks
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 9 | 8
score on a scale | -21.3 (33.88) | 10.4 (31.10)

18. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 29 weeks
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 4 | 5
score on a scale | -12.5 (35.03) | 5.0 (18.26)

19. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 41 weeks
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 2 | 2
score on a scale | 8.3 (11.79) | -16.7 (23.57)

20. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 54 weeks
Population: Due to the premature termination of the study, there was insufficient data to allow statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 1 | 1
score on a scale | -8.3 (NA) — Only 1 patient so no SD | -33.3 (NA) — Only 1 patient so no SD

21. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 66 weeks
Population: No data collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Health-related Quality of Life on the 4- and 7-point EORTC QLQ-C30
Description: as for outcome 14
Time Frame: Baseline, 78 weeks
Population: No data collected
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 26 months
Description: The SMC alone group enrolled 13 subjects but only 10 were treated thus there were only 10 subjects at risk for adverse events.
Arm/Group | Photodynamic Therapy-Photofrin Plus SMC | Standard Medical Care (SMC)
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 11/15 | 10/10
Other Adverse Events (participants affected / at risk) | 13/15 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy-Photofrin Plus SMC (N=15) | Standard Medical Care (SMC) (N=10)
Sepsis (Infections and infestations) | 5 (8) | 3 (4)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Liver abcess (Infections and infestations) | 1 (1) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 6 (6) | 9 (9)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Post-procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy-Photofrin Plus SMC (N=15) | Standard Medical Care (SMC) (N=10)
Nausea (Gastrointestinal disorders) | 9 (9) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (6) | 2 (4)
Pyrexia (General disorders) | 3 (3) | 6 (6)
Chills (General disorders) | 4 (4) | 4 (4)
Asthenia (General disorders) | 3 (3) | 2 (2)
Catheter site pain (General disorders) | 2 (2) | 1 (1)
Edema peripheral (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hypokaliemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Iron deficiency anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bilirubine increase (Investigations) | 3 (3) | 0 (0)
CA-19 increase (Investigations) | 2 (2) | 0 (0)
GGT (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Uretherolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Nausea (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Skin cut (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Aplastic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjuctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feces discolored (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Catheter site discharge (General disorders) | 1 (1) | 1 (1)
Catheter site injury (General disorders) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Influenza-like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary tract infection bacteria (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Hemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Pulse abnormal (Investigations) | 1 (1) | 0 (0)
Fluid imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkaliemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamine D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asterixis (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Food aversion (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Urethrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythmetous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated due to low accrual. Consequently, there was insufficient data to allow statistical analysis. Only descriptive statistics are presented for the primary endpoint, overall survival time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less